CLINICAL TRIAL: NCT02714088
Title: The Effect of Novel High-intensity Interval Training on Physical Fitness in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Christopher Hurst, Postgraduate Researcher, Teesside University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TEES-CH170216-SSSBL
Record Dates: First submitted 2016-03-08; First posted 2016-03-21 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: High-intensity Interval Training
Keywords: High-intensity interval training; Functional fitness; Quality of life; Older adults

ARMS (2):
- Intervention (Experimental): Participants will undertake a high-intensity interval training intervention, completing two exercise sessions per week for 12 weeks. The exercise sessions will consist of 4 sets of 4-6 repetitions of 60s (45s high-intensity exercise, followed by 15s rest), interspersed with 3 minutes rest. During each exercise repetition participants will be encouraged to reach >90% of their maximal heart rate.
  Interventions: Other: Novel high-intensity interval training
- Control (No Intervention): Participants will not undertake any formal intervention and will be asked to maintain their usual physical activity habits and diet.

INTERVENTIONS:
Other: Novel high-intensity interval training
  Arms: Intervention

SUMMARY:
High-intensity interval training (HIT) has been demonstrated to be an effective strategy to improve markers of health and fitness across a wide range of healthy and clinical populations. Currently however, there is only limited evidence which has examined the effectiveness of HIT in older adults (>50 years). HIT is an appealing strategy in this group as it has the potential to impact both cardiorespiratory and muscular fitness, which both play an important role in maintaining functional fitness and quality of life in a time-efficient manner. Developing an understanding of novel strategies for delivering this type of exercise training may ultimately provide a viable alternative to traditional modes of exercise training for a broader range of participants. As such, the purpose of this study is to evaluate the effects of a novel, high-intensity interval training exercise protocol to improve physical fitness in adults aged over 50 years. This research also aims to evaluate if this type of training intervention is feasible in this population, through analysis of adherence and intervention fidelity.

ELIGIBILITY:
Inclusion Criteria:

1. Must be aged 50-85 years
2. Must be able to provide informed consent to participate
3. Must be free from all exclusion criteria

Exclusion Criteria:

1. Symptoms of or known presence of heart disease of major atherosclerotic cardiovascular disease
2. Early family history of sudden cardiac death
3. Condition or injury or co-morbidity affecting the ability to undertake exercise
4. Diabetes mellitus
5. Pregnancy or likelihood of pregnancy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in lower body muscular power | Baseline and following exercise training (12 weeks)
  Assessed via Nottingham Leg Extensor Power Rig
Change in Aerobic fitness | Baseline and following exercise training (12 weeks)
  Assessed via Chester step test
Change in upper extremity muscular strength | Baseline and following exercise training (12 weeks)
  Hand grip strength assessed using handheld dynamometer
Change in quality of life | Baseline and following exercise training (12 weeks)
  Assessed via Short form quality of life questionnaire (SF36)

OTHER OUTCOMES:
Heart rate during high-intensity interval training exercise sessions | Up to 12 weeks
Rating of perceived exertion (RPE) during high-intensity interval training exercise sessions | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Teesside University, Middlesbrough, Tees Valley, United Kingdom